CLINICAL TRIAL: NCT04223375
Title: Effect of Nutrition Training on Mother's Nutrition Pattern, Breast Milk and Newborn Intestinal Microbiota
Brief Title: Effect of Nutrition Training on Mothers' Nutrition Pattern, Breast Milk and Newborn Intestinal Microbiota
Acronym: microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, gnacar, Effect of Nutrition Training on Mothers' Nutrition Pattern, Breast Milk and Newborn Intestinal Microbiota, Inonu University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Turgut Özal
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Microbial Colonization; Nutrient Deficiency
Keywords: microbiata; food groups
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Group (Experimental): After the health status of the mothers in the experimental group was stabilized, approximately 20-30 minutes of nutritional education was given at the first interview before the hospital discharge. After nutrition education, motivational messages were sent to women's phones once a week. In addition, mothers were given nutritional counseling during their home visits during the 1st and 3rd months, and their questions and problems regarding nutrition were evaluated. The mother was supported where she needed it.
  In nutritional education, information was given such as adequate and balanced nutrition in the postpartum period, adequate fluid intake, consumption and importance of prebiotic and probiotic foods, the importance of healthy microbiota for infant health and the amount of nutrients equivalent to one serving. In addition, the handbook which contains the educational content is given to the mothers to facilitate the recall.
  Interventions: Behavioral: Nutrition Training
- Control Group (No Intervention): No intervention was made to the control group.

INTERVENTIONS:
Behavioral: Nutrition Training — Postpartum women were educated on postpartum healthy and regular nutrition.
  Arms: Nutrition Group

SUMMARY:
Objective: The aim of this study was to investigate the effects of nutrition Training on mothers' nutrition pattern, breast milk and newborn intestinal microbiota.

Materials and methods: The study was conducted as a non-randomized controlled experimental study. The population of the study consisted of mothers and their babies who delivered vaginally, breastfeeded their babies at the end of the second postnatal day and delivered at the maternity ward of the Malatya Training and Research Hospital Beydağı Campus. The sample of the study consisted of 120 mothers, 57 of whom were experimental and 63 of them were in the control group. In this study, a sub-sample of 15 mothers and their infants was selected and microbiota of breast milk and stool samples were examined.

In the first interview with the mothers in the experimental and control groups, Participant Identification Form, BTSKF were applied as a pre-test and stool samples of breast milk and newborn were taken. Then, the mothers in the experimental group were given nutritional education. In addition, motivational messages were sent to mothers' phones once a week. MTS in the experimental and control groups were filled with BTSKF as an intermediate test at the first month and post-test at the third month and stool samples of breast milk and newborn were collected at the mothers' own homes. During these visits, nutrition counseling was given to the mothers in the experimental group.

DETAILED DESCRIPTION:
Nutrition is very important from intrauterine life to old age for a healthy and productive life. However, the importance of pregnancy, childbirth and breastfeeding during the special stages in which the woman is experienced in her life process increases slightly (Ho et al., 2016; Erick, 2018; Tekiner and Ungan, 2014). Healthy nutrition is a key concern for the health of the baby during pregnancy, childbirth and breastfeeding periods as well as the health of the mother (Taşkın, 2016; Samur, 2008). Intrauterine life is transmitted by placental way and in the postpartum period, breast milk is fed to the baby. Therefore, in order to ensure optimal growth and development of the baby, the mother needs adequate, regular and quality nutrition (Ho et al., 2016; Erick, 2018; Tekiner and Ungan, 2014).

ELIGIBILITY:
Inclusion Criteria:

* Being literate,
* Being within 48 hours after delivery,
* No disease / complications in mother and newborn,
* Delivery at term (according to the first day of the last menstrual period).

Exclusion Criteria:

• A mother's inability to breastfeed her baby for a variety of reasons, either short or long term (mastitis, abscess).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Effect of nutrition traning | 3 months
  Food Consumption Frequency Registration Form It is a form created by determining the type, frequency and amount of food consumed in order to determine the food consumption habits of mothers in the last 1 month. Food Consumption Frequency Registration Form is composed of four basic food groups (Milk and dairy products,Meat and group foods, Vegetable and fruit group and Grain group).
  Mothers were asked to define the frequency of food consumption as daily, 5-6 times a week, 3-4 times a week, 1-2 times a week, once every 15 days and once a month. The mother of the amount of food they consume is used in everyday life, cups, spoons, were asked to specify the dimensions such as grain, followed by Turkey Ministry of Health Nutrition Guidelines (2016) was recorded by turning a portion.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin NACAR, Msc, Study Director — Inonu University
Locations (1):
- Inonu University, Malatya, Battalgazi, Turkey (Türkiye)

REFERENCES:
- [Background] Timur Tashan S, Ucar T, Aksoy Derya Y, Nacar G, Erci B. Validity and Reliability of the Turkish Version of the Modified Breast Cancer Worry Scale. Iran J Public Health. 2018 Nov;47(11):1681-1687. PMID 30581784
- See also: Validity and Reliability of the Turkish Version of the Modified Breast Cancer Worry Scale. — http://www.ncbi.nlm.nih.gov/pubmed/30581784